CLINICAL TRIAL: NCT00828165
Title: A Safety Study of ARRY-300 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: ARRAY-300-101
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARRY-300 (Experimental)
  Interventions: Drug: ARRY-300, MEK inhibitor; oral
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARRY-300, MEK inhibitor; oral — single dose, escalating
  Arms: ARRY-300
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1 study, involving a 1-day dosing period (up to 3 dosing periods per subject), designed to test the safety of investigational study drug ARRY-300 in healthy subjects. Approximately 12 healthy subjects from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male or female (females must be of non-childbearing potential) between the ages of 18 and 50 years, inclusive.
* Body mass index (BMI) of 18 kg/m2 to 35 kg/m2; and a total body weight > 50 kg (110 lbs) and < 113 kg (280 lbs).
* Additional criteria exist.

Key Exclusion Criteria:

* Evidence or history of clinically significant hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, dermatologic, or allergic disease (including drug allergies that are clinically significant and not remote, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* A condition possibly affecting drug absorption (e.g., gastrectomy).
* Women who are pregnant or breastfeeding.
* A positive test for drugs or alcohol.
* Use of tobacco- or nicotine-containing products in excess of 5 cigarettes per day, or daily use of pipe, cigar, chewing tobacco or nicotine gum or patches.
* Treatment with an investigational drug within 30 days prior to first dose of study drug.
* Use of prescription or nonprescription drugs, vitamins, grapefruit juice, and dietary or herbal supplements within 14 days prior to the first dose of study drug. As exceptions, acetaminophen may be used at doses of ≤ 1 g/day or ibuprofen may be used at doses of ≤ 800 mg/day until 24 hours prior to first dose of study drug.
* Blood donation of ≥ 1 pint within 30 days prior to first dose of study drug.
* Evidence of hepatitis B or C, or human immunodeficiency virus (HIV) infection upon serological testing.
* Additional criteria exist.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, vital signs and electrocardiograms. | Duration of study
Characterize the pharmacokinetics (PK) of the study drug and metabolites in terms of plasma concentrations. | Following a single dose

SECONDARY OUTCOMES:
Characterize the pharmacodynamic (PD) activity of the study drug on biomarkers. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- PPD Development, LP, Austin, Texas, United States